CLINICAL TRIAL: NCT05587868
Title: Karakteristik Dan Pengaruh Vaksinasi COVID-19 Terhadap Klinis Dan Kualitas Hidup Pasien Long COVID di RSUPN Dr. Cipto Mangunkusumo
Brief Title: COVID-19 Vaccination Status and The Clinical Outcomes of Long COVID-19 Patients
Acronym: SURVIVOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Eric Daniel Tenda MD, DIC, PhD, Academic Staff in Respirology and Critical Illness Division, Department of Internal Medicine, Dr. Cipto Mangunkusumo General Hospital, Jakarta, Indonesia, Indonesia University
Other Study IDs: 21-10-1101
Record Dates: First submitted 2022-10-19; First posted 2022-10-20 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; SARS CoV-2 Infection
Keywords: Long COVID; Post COVID-19 Syndrome; Post-Acute Sequelae of SARS-CoV2 Infection (PASC); Chronic COVID-19; Post-Acute COVID-19; Long-haulers; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients who have not received vaccination for COVID-19: This group includes patients who refused or contraindicated to receive vaccination for COVID-19.
- Patients who had received first dose of vaccination for COVID-19: Regardless of the type of COVID-19 vaccine used (received before or after laboratory-confirmed SARS-CoV-2 infection).
  Interventions: Biological: COVID-19 Vaccine
- Patients who had received second dose vaccination for COVID-19: Regardless of the type of COVID-19 vaccine used, using same type of vaccine as the first dose (received before and/or after laboratory-confirmed SARS-CoV-2 infection).
  Interventions: Biological: COVID-19 Vaccine
- Patients who had received third dose/booster vaccination for COVID-19: Complete cycle of vaccination using same type of vaccine for the first and second dose and a same/different type for the third dose/booster (received before and/or after laboratory-confirmed SARS-CoV-2 infection).
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Mandatory COVID-19 vaccination as part of the the Indonesian national government program.
  Groups: Patients who had received first dose of vaccination for COVID-19; Patients who had received second dose vaccination for COVID-19; Patients who had received third dose/booster vaccination for COVID-19

SUMMARY:
Long COVID is defined by the persistence or emergence of symptoms for more than 4 weeks beyond the acute phase of Severe Acute Respiratory Syndrome-Corona Virus-2 (SARS-CoV-2) infection. As the number of cases increases and various strains of SARS-CoV-2 emerge, so does the number of long COVID cases. Various multi-organ complications after COVID-19 infection include respiratory, cardiovascular, gastrointestinal, hepatobiliary, metabolic, and neuropsychiatric disorders. The symptoms and characteristics of Long COVID vary in each country.

Vaccination against SARS-CoV-2 has been documented to increase clinical resolution of Long COVID. In Indonesia, current full-dose vaccination coverage had merely reached 15.6% of the national vaccination target. This condition can be predictably associated with a longer duration and higher severity of symptoms in Long COVID patients.

The purpose of this study is to provide an overview of the symptoms and characteristics and determine whether vaccination against SARS-CoV-2 could improve clinical outcomes and quality of life of Long COVID patients at Dr. Cipto Mangunkusumo General Hospital.

DETAILED DESCRIPTION:
The study is a prospective cohort study designed to assess whether vaccination against SARS-CoV-2 could reduce the severity and duration of Long COVID, resulting in changes in quality of life in Long-COVID patients. This study was approved by the Institutional Review Board of Universitas Indonesia and informed consent was obtained before enrollment for patients eligible for this study. Allocation of participants to each group was done via vaccination status data collected before enrollment in this study.

Baseline participant characteristics were collected before enrollment, including age, sex, body mass index, alcohol and smoking consumption, comorbidities, documented vaccination status, detailed history of laboratory-confirmed SARS-CoV-2 infection, Long COVID symptoms, severity, and duration. The Six-Minute Walking Test (6MWT) was performed according to the guidelines of the American Thoracic Society (ATS) to assess functional exercise capacity in each patient, followed by a quality of life assessment using the St George's Respiratory Questionnaire (SGRQ) and the Short Form (SF)-36 Health Survey questionnaire.

The primary outcomes of this study were long-COVID patients' characteristics, symptom phenotype, and changes in quality of life. The investigators anticipated a change in quality of life difference of 20%, with statistical power of 80% and a level of significance of 0.05. The total required sample size was 192 participants. In anticipation of participant drop-out, the investigators planned to recruit a total of 250 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥ 18 years
2. History of laboratory-confirmed SARS-CoV-2 infection via a positive molecular (RT-PCR) or antigen (lateral flow assay) test, receiving outpatient/inpatient care from Dr. Cipto Mangunkusumo General Hospital, anytime prior to enrollment in this study
3. Patients with/without comorbidities
4. Willing to fill-out online Long COVID symptoms follow-up questionnaire
5. Willing and able to comply with trial protocol (re-visits and physical testing)

Exclusion Criteria:

1. Patients with no registered medical record number (MRN) at Dr. Cipto Mangunkusumo General Hospital
2. Refusal to participate in the study or to sign the informed consent form
3. Any contraindications for 6 Minute Walking Test according to the guidelines of the American Thoracic Society (ATS)
4. Patients with no access to a smartphone or computer (desktop, laptop, or tablet) to fill out the online screening questionnaire
5. Patients who died during or before enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long COVID-19 patients received outpatient/inpatient care from Dr. Cipto Mangunkusumo General Hospital during the COVID-19 infection anytime before enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Long COVID symptoms phenotype | Up to 6 months
  Wide range of symptoms associated with Long COVID in which people have persistent or emerging symptoms > 4 weeks after an initial SARS-CoV-2 infection.
  In this study symptoms will be reported and analyzed by both symptom clusters and individual symptoms.
Change in quality of life (QoL), self-assessed using the St George's Respiratory Questionnaire (SGRQ) | Baseline, 3 and 6 months
  SGRQ addresses QoL in the domains of symptoms, activity, impacts within last 4 weeks. Symptoms, activity, impacts and total score are calculated to summarises the impacts of the disease on overall health status. Total score ranges from 100 (worst possible health status) to 0 (best possible health status).
Change in quality of life (QoL), self-assessed using the Short Form (SF)-36 Health Survey questionnaire | Baseline, 3 and 6 months
  SF-36 Health Survey questionnaire addresses QoL in the domains of vitality, physical functioning, bodily pain, general health perceptions, physical and emotional and social role functioning. The final score ranges from 0 (worse health status) to 100 (better health status).

SECONDARY OUTCOMES:
Change in functional exercise capacity, objectively measured using Six-Minute Walking Test (6MWT) | Baseline, 3 and 6 months
  Performed according to the guidelines of American Thoracic Society (ATS)
  6MWT evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism.
  During the 6MWT, such data are collected:
  * Pre-post test: blood pressure, oxygen saturation (SpO2), heart rate, dyspnea and overall fatigue score using the Modified Borg scale
  * One time measurement: total distance walked in 6 minutes, symptoms at the end of exercise
Change in symptoms severity | Baseline, 3 and 6 months
  Subjectively measured using online self-assessed symptoms follow-up questionnaire, disease severity is measured using ordinal scale, with 11 steps ranging from 0 (no symptoms) to 10 (Very severe).
  The change in symptom severity will be described by whether participants report that symptoms have become more severe, less severe, or did not change severity.
Change in symptoms frequency | Baseline, 3 and 6 months
  Subjectively measured using online self-assessed symptoms follow-up questionnaire, symptom frequency is measured using ordinal scale, with 11 steps ranging from 0 (no symptoms) to 10 (All time).
  The study outcome will be reported by both symptom clusters and individual symptoms. The change in symptom frequency will be described by whether participants report that symptoms have become more frequent, less frequent, or did not change.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Tenda, MD, DIC, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia - Dr Cipto Mangunkusumo General Hospital
Locations (1):
- Respirology and Critical Care Medicine Division, Departement of Internal Medicine, Dr Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Chopra V, Flanders SA, O'Malley M, Malani AN, Prescott HC. Sixty-Day Outcomes Among Patients Hospitalized With COVID-19. Ann Intern Med. 2021 Apr;174(4):576-578. doi: 10.7326/M20-5661. Epub 2020 Nov 11. No abstract available. PMID 33175566
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Arnold DT, Milne A, Samms E, Stadon L, Maskell NA, Hamilton FW. Are Vaccines Safe in Patients with Long COVID? A prospective Observational Study. medRxiv. 2021; 03.11.21253225
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Gupta A, Madhavan MV, Sehgal K, Nair N, Mahajan S, Sehrawat TS, Bikdeli B, Ahluwalia N, Ausiello JC, Wan EY, Freedberg DE, Kirtane AJ, Parikh SA, Maurer MS, Nordvig AS, Accili D, Bathon JM, Mohan S, Bauer KA, Leon MB, Krumholz HM, Uriel N, Mehra MR, Elkind MSV, Stone GW, Schwartz A, Ho DD, Bilezikian JP, Landry DW. Extrapulmonary manifestations of COVID-19. Nat Med. 2020 Jul;26(7):1017-1032. doi: 10.1038/s41591-020-0968-3. Epub 2020 Jul 10. PMID 32651579
- [Background] Garrigues E, Janvier P, Kherabi Y, Le Bot A, Hamon A, Gouze H, Doucet L, Berkani S, Oliosi E, Mallart E, Corre F, Zarrouk V, Moyer JD, Galy A, Honsel V, Fantin B, Nguyen Y. Post-discharge persistent symptoms and health-related quality of life after hospitalization for COVID-19. J Infect. 2020 Dec;81(6):e4-e6. doi: 10.1016/j.jinf.2020.08.029. Epub 2020 Aug 25. PMID 32853602
- [Background] Shang J, Ye G, Shi K, Wan Y, Luo C, Aihara H, Geng Q, Auerbach A, Li F. Structural basis of receptor recognition by SARS-CoV-2. Nature. 2020 May;581(7807):221-224. doi: 10.1038/s41586-020-2179-y. Epub 2020 Mar 30. PMID 32225175
- [Background] Goertz YMJ, Van Herck M, Delbressine JM, Vaes AW, Meys R, Machado FVC, Houben-Wilke S, Burtin C, Posthuma R, Franssen FME, van Loon N, Hajian B, Spies Y, Vijlbrief H, van 't Hul AJ, Janssen DJA, Spruit MA. Persistent symptoms 3 months after a SARS-CoV-2 infection: the post-COVID-19 syndrome? ERJ Open Res. 2020 Oct 26;6(4):00542-2020. doi: 10.1183/23120541.00542-2020. eCollection 2020 Oct. PMID 33257910
- [Background] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Background] Lopez-Leon S, Wegman-Ostrosky T, Perelman C, Sepulveda R, Rebolledo PA, Cuapio A, Villapol S. More than 50 Long-term effects of COVID-19: a systematic review and meta-analysis. medRxiv [Preprint]. 2021 Jan 30:2021.01.27.21250617. doi: 10.1101/2021.01.27.21250617. PMID 33532785
- [Background] Udwadia ZF, Koul PA, Richeldi L. Post-COVID lung fibrosis: The tsunami that will follow the earthquake. Lung India. 2021 Mar;38(Supplement):S41-S47. doi: 10.4103/lungindia.lungindia_818_20. PMID 33686978
- [Background] Wang Y, Dong C, Hu Y, Li C, Ren Q, Zhang X, Shi H, Zhou M. Temporal Changes of CT Findings in 90 Patients with COVID-19 Pneumonia: A Longitudinal Study. Radiology. 2020 Aug;296(2):E55-E64. doi: 10.1148/radiol.2020200843. Epub 2020 Mar 19. PMID 32191587
- [Background] Mo X, Jian W, Su Z, Chen M, Peng H, Peng P, Lei C, Chen R, Zhong N, Li S. Abnormal pulmonary function in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jun 18;55(6):2001217. doi: 10.1183/13993003.01217-2020. Print 2020 Jun. PMID 32381497
- [Background] Inciardi RM, Lupi L, Zaccone G, Italia L, Raffo M, Tomasoni D, Cani DS, Cerini M, Farina D, Gavazzi E, Maroldi R, Adamo M, Ammirati E, Sinagra G, Lombardi CM, Metra M. Cardiac Involvement in a Patient With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):819-824. doi: 10.1001/jamacardio.2020.1096. PMID 32219357
- [Background] Huang L, Zhao P, Tang D, Zhu T, Han R, Zhan C, Liu W, Zeng H, Tao Q, Xia L. Cardiac Involvement in Patients Recovered From COVID-2019 Identified Using Magnetic Resonance Imaging. JACC Cardiovasc Imaging. 2020 Nov;13(11):2330-2339. doi: 10.1016/j.jcmg.2020.05.004. Epub 2020 May 12. PMID 32763118
- [Background] McMahon DE, Gallman AE, Hruza GJ, Rosenbach M, Lipoff JB, Desai SR, French LE, Lim H, Cyster JG, Fox LP, Fassett MS, Freeman EE. Long COVID in the skin: a registry analysis of COVID-19 dermatological duration. Lancet Infect Dis. 2021 Mar;21(3):313-314. doi: 10.1016/S1473-3099(20)30986-5. Epub 2021 Jan 15. No abstract available. PMID 33460566
- [Background] Mehta P, Bunker CB, Ciurtin C, Porter JC, Chambers RC, Papdopoulou C, Garthwaite H, Hillman T, Heightman M, Howell KJ, Eleftheriou D, Denton CP. Chilblain-like acral lesions in long COVID-19: management and implications for understanding microangiopathy. Lancet Infect Dis. 2021 Jul;21(7):912. doi: 10.1016/S1473-3099(21)00133-X. Epub 2021 Mar 8. No abstract available. PMID 33705725
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Stefano GB, Ptacek R, Ptackova H, Martin A, Kream RM. Selective Neuronal Mitochondrial Targeting in SARS-CoV-2 Infection Affects Cognitive Processes to Induce 'Brain Fog' and Results in Behavioral Changes that Favor Viral Survival. Med Sci Monit. 2021 Jan 25;27:e930886. doi: 10.12659/MSM.930886. PMID 33487628
- [Background] Parker AM, Sricharoenchai T, Raparla S, Schneck KW, Bienvenu OJ, Needham DM. Posttraumatic stress disorder in critical illness survivors: a metaanalysis. Crit Care Med. 2015 May;43(5):1121-9. doi: 10.1097/CCM.0000000000000882. PMID 25654178
- [Background] Nikayin S, Rabiee A, Hashem MD, Huang M, Bienvenu OJ, Turnbull AE, Needham DM. Anxiety symptoms in survivors of critical illness: a systematic review and meta-analysis. Gen Hosp Psychiatry. 2016 Nov-Dec;43:23-29. doi: 10.1016/j.genhosppsych.2016.08.005. Epub 2016 Aug 28. PMID 27796253
- [Background] Sansone A, Mollaioli D, Ciocca G, Limoncin E, Colonnello E, Vena W, Jannini EA. Addressing male sexual and reproductive health in the wake of COVID-19 outbreak. J Endocrinol Invest. 2021 Feb;44(2):223-231. doi: 10.1007/s40618-020-01350-1. Epub 2020 Jul 13. PMID 32661947
- See also: WHO Coronavirus (COVID-19) - Dashboard — https://covid19.who.int
- See also: Long COVID: the NHS plan for 2021/22 — https://england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2021/06/C1312-long-covid-plan-june-2021.pdf

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT05587868/Prot_SAP_ICF_000.pdf